CLINICAL TRIAL: NCT05284721
Title: A Family Peer Navigator Model to Increase Access and Initial Engagement in Coordinated Specialty Care Programs Among Black Families
Brief Title: Family Peer Navigator for Early Psychosis for Black Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Oladunni Oluwoye, Assistant Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19181-001
Record Dates: First submitted 2022-02-28; First posted 2022-03-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Family Members
Keywords: Black/African American; Early Psychosis; Access and Engagement
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care Coordination Phase III (Active Comparator): Family member participants randomized to the active control will receive two brief psychoeducation sessions, two brief check ins across one month and linked to appropriate services.
  Interventions: Behavioral: Care Coordination
- Family Peer Navigator model Psychosis Phase III (Experimental): Family member participants randomized to the Family Peer Navigator condition will participate in two sessions for introduction/assessment, four individual psychoeducation sessions, and six brief check ins delivered by Family Peer Navigators.
  Interventions: Behavioral: Family Peer Navigator for Early Psychosis

INTERVENTIONS:
Behavioral: Family Peer Navigator for Early Psychosis — The Family Peer Navigator model is theoretical underpinning by the Social-Ecological Model and the Social Cognitive Theory, that incorporates a mixture of evidence- and research-based strategies, to include three key components: 1) Introduction and Assessment; 2) Individual Psychoeducation; 3) Six Brief Check-In
  Arms: Family Peer Navigator model Psychosis Phase III
Behavioral: Care Coordination — active control, treatment as usual including services provided by the coordinated specialty care program for first-episode psychosis.
  Arms: Care Coordination Phase III

SUMMARY:
Building upon formative research, this mixed methods study will be conducted in three phases to develop, refine, and pilot-test a multi-component Family Peer Navigator model designed to increase access to and initial engagement in coordinated specialty care for early psychosis among Black/African American families.

DETAILED DESCRIPTION:
The overall goal of this mixed methods study will be conducted in three phases to develop, refine, and pilot-test a multi-component Family Peer Navigator model designed to increase access to and engagement in coordinated specialty care programs among Black/African American families. Phase II will recruit 10 family member participants to complete a four-month open trial to refine the Family Peer Navigator model. During Phase III, a total of 40 Black/African American families will be recruited to participate in a randomized pilot trial of the Family Peer Navigator model against a low-intensive care coordination in two coordinated specialty care programs to assess acceptability, feasibility, and preliminary impact.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Identifies as Black/African American
3. Loved one who meets criteria for risk of psychosis with a total score of ≥ 3 on the Prodromal Questionnaire- Brief Version

Exclusion Criteria:

1. Family members who cannot understand the consent process
2. Non-English speaking adults
3. Black/African American families referred to coordinated specialty care and who have already been determined eligible for services by providers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire-8 (CSQ-8) | Months 1 through 3 of treatment period; repeated measure to assess change in acceptability through study completion, average of 4 months
  Self-report measure to assess acceptability, a brief measure for family member participant. Items are scored from 1 to 4. Possible total scores range from 8 to 32, with higher scores (>23) indicating greater satisfaction.
Youth Services Survey-Families (YSS-F) | Baseline and Month 3 of treatment period; repeated measure to assess change in acceptability through study completion, average of 4 months
  Self-report measure to assess acceptability in the following domains: appropriateness, participation, cultural sensitivity, social connectedness, and outcomes. Items in a domain are summed and divided by the total number of items, and scores greater than 3.5 are reported in the positive range for the domain.
Number of Referrals (Recruitment) to assess feasibility | Baseline through study completion; repeated measure to assess change in feasibility through study completion, average of 4 months
  The number of family member participants recruited and referrals received categorized by where they originated.
Level of Engagement to measure feasibility | Baseline through study completion; repeated measure to assess change in feasibility through study completion, average of 4 months
  Total number of sessions attended, the number of contact hours with families and by which method (videoconference, in person, text, email etc.) and the number of completed measures.
Rate of Retention to measure feasibility | Baseline through study completion; repeated measure to assess change in feasibility through study completion, average of 4 months
  The percentage of families that drop out (family declined or missed 3 consecutive appointments).

SECONDARY OUTCOMES:
General Self-Efficacy scale | Baseline through study completion; repeated measure to assess change through study completion, average of 4 months
  A self report measure of self-efficacy correlated to emotion, optimism and work satisfaction. Scores range from 10 to 40 with higher scores indicating more self-efficacy.
Youth Services Survey for Families - Social Connectedness Subscale | Baseline through study completion; repeated measure to assess change through study completion, average of 4 months
  Social connectedness will be measured using four questions (e.g., "I know people who will listen and understand me when I need to talk") from the YSS-F. Scores range from 4 to 20, higher scores indicating greater social connectedness.
Culturally-adapted Knowledge about Psychosis questionnaire (CaKAP) | Baseline through study completion; repeated measure to assess change through study completion, average of 4 months
  Self-reported measure that includes 23 culturally specific items across five subscales: symptoms and problems relating to psychosis; cause; other treatments and services; course and outcome; and management. Total scores range from 0 through 104 where higher scores indicate greater knowledge.
Youth Services Survey for Families - Cultural Sensitivity Subscale | Baseline through study completion; repeated measure to assess change through study completion, average of 4 months
Scale to Assess Therapeutic Relationships in Community Mental Health Care (STAR) | Baseline through study completion; repeated measure to assess change through study completion, average of 4 months
  Measure includes 12-items to assess therapeutic relationships.

OTHER OUTCOMES:
Time from Referral to Enrollment to assess | Baseline through study completion, average of 4 months
  Provider reported measure used to assess the access to coordinated specialty care programs which a participant had as defined as the time between point of referral to receipt of mental health service.
Initial Engagement to assess preliminary effectiveness | Baseline through study completion, average of 4 months
  Provider reported measure defined as >1 attendance or contact for the family appointment within 30 days of loved ones' intake in mental health program.
Adherence to model | Baseline through study completion; repeated measure to assess the implementation feasibility of services through study completion, average of 4 months
  Feasibility checklists to measure the amount and percentage of components delivered. A structured meeting log will be maintained by study staff to document solutions, barriers and challenges to implementation as well as the number of meetings scheduled and attended.

CONTACTS AND LOCATIONS:
Locations (1):
- New Journeys: Coordinated Specialty care, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oluwoye O, Stokes BI, Burduli E, Kriegel LS, Hoagwood KE. Community-based family peer navigator programme to facilitate linkage to coordinated specialty care for early psychosis among Black families in the USA: A protocol for a hybrid type I feasibility study. BMJ Open. 2023 Jul 5;13(7):e075729. doi: 10.1136/bmjopen-2023-075729. PMID 37407058